CLINICAL TRIAL: NCT05776277
Title: A Two-stage, Randomized, Controlled Trial Comparing the Safety and Efficacy of Iltamiocel With Placebo in the Treatment of Female Participants With Chronic Fecal Incontinence and a History of Obstetric Anal Sphincter Injury (DigniFI)
Brief Title: Iltamiocel Compared to Placebo for Chronic Fecal Incontinence in Females With Obstetric Injury
Acronym: DigniFI
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Cook MyoSite (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 22-01
Record Dates: First submitted 2023-03-08; First posted 2023-03-20 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Fecal Incontinence
Keywords: Obstetric Trauma; Obstetric Injury; Cell Therapy; Anal Incontinence; Rectal Diseases; Intestinal Diseases; Gastrointestinal Diseases; Bowel Incontinence
MeSH Terms: conditions — Fecal Incontinence; Encopresis; Rectal Diseases; Intestinal Diseases; Gastrointestinal Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Iltamiocel (Experimental)
  Interventions: Biological: Iltamiocel
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Iltamiocel — Single external anal sphincter (EAS) injection of 300 x 10^6 cells.
  Arms: Iltamiocel
Other: Placebo — Placebo control is the vehicle solution used for the study product.
  Arms: Placebo

SUMMARY:
This study evaluates the efficacy and safety of a single injection of iltamiocel (300 x 10^6 cells) compared to a placebo in the reduction of fecal incontinence episode frequency in adult female participants with chronic fecal incontinence and a history of obstetric anal sphincter injury. Half of the participants will receive iltamiocel (injections with cells) and the other half will receive placebo.

DETAILED DESCRIPTION:
Chronic fecal incontinence (FI) is the recurrent unintended passage of mucus and/or liquid or solid stool for at least 6 months. Iltamiocel is an investigational cell therapy product that involves a medical procedure in which a participant's own muscle cells are collected, processed, and then injected into the tissues of the external anal sphincter.

This is a double-blind randomized study, which means neither the participant, nor the study doctor will know which treatment group the participant will be in. Participants who are randomly chosen to receive injection with placebo will have the option to receive an injection with their cells after completion of the blinded portion of their study participation (12 months).

ELIGIBILITY:
Inclusion Criteria:

* Adult female ≥ 18 years of age who has primary symptoms of fecal incontinence (FI) for at least 12 months.
* History of obstetric anal sphincter injury (e.g., episiotomy, perineal tear).
* Failed conservative treatment (e.g., dietary modification, antidiarrheal medications, pelvic floor muscle training, biofeedback) for at least 6 months prior to enrollment.
* Must be willing and able to comply with the study procedures, be mentally competent and able to understand all study requirements, and must agree to read and sign the informed consent form prior to any study-related procedures.

Exclusion Criteria:

* Has an implanted stimulation neuromodulation system (sacral or tibial) and symptoms are unstable as determined by the physician.
* Is pregnant or planning to become pregnant within the next 2 years.
* Has known rectal sensory dysfunction (e.g., hypersensitivity or hyposensitivity).
* Has an obstetric anal sphincter injury (e.g., episiotomy, perineal tear) within 1 year previous to study enrollment.
* Patient BMI ≥ 38.
* Has a history of cancer in the colorectal or pelvic organs within 5 years prior to study enrollment.
* Any cancer that has undergone treatment within the past 12 months.
* Has an established diagnosis of inflammatory bowel disease (Crohn's disease, ulcerative colitis) or current intestinal stoma.
* Has grade III/IV hemorrhoids.
* Has chronic diarrhea at the time of Screening.
* Has chronic constipation at the time of Screening.
* Has significant pelvic floor prolapse, significant genitourinary prolapse beyond the introitus, significant symptomatic rectocele, or evidence of significant rectal evacuation disorder leading to post-defecatory leakage.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-03-21 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Changes in frequency of fecal incontinence episodes. | 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Ron Jankowski, PhD, Study Director — Cook Myosite, Inc.
Locations (25):
- United States (25):
  - UC San Diego Health, La Jolla, California
  - UC Irvine Medical Center, Orange, California
  - University of California, San Francisco - Center for Colorectal Surgery, San Francisco, California
  - Prestige Medical Group, Tustin, California
  - American Association of Female Pelvic Medicine, Westlake Village, California
  - University of Florida Shands Hospital, Gainesville, Florida
  - Healthcare Clinical Data, Inc., Miami, Florida
  - Orlando Health Colon & Rectal Institute, Orlando, Florida
  - USF Health South Tampa Center for Advanced Healthcare, Tampa, Florida
  - Colorectal Wellness Center, Fayetteville, Georgia
  - University of Illinois, Chicago, Illinois
  - Franciscan Health Indianapolis, Indianapolis, Indiana
  - Ochsner Health, New Orleans, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Bennett Institute of Urogynecology and Incontinence, Grand Rapids, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Rutgers, Robert Wood Johnson Medical School, Clinical Research Center, New Brunswick, New Jersey
  - Westchester Medical Center, Hawthorne, New York
  - The Mount Sinai Medical Center, New York, New York
  - Weill Cornell Medicine, New York, New York
  - Stony Brook University Hospital, Stony Brook, New York
  - Cleveland Clinic Main Campus Crile Building, Cleveland, Ohio
  - Rhode Island Hospital, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: No